CLINICAL TRIAL: NCT00005342
Title: Weight Set-Point and HDL Concentration in Runners
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4205; R01HL045652 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2000-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To investigate the differences in diet, fat cell morphology and lipoprotein metabolism in previously- overweight and naturally lean men and women who ran and who lived sedentary lifestyles in order to better understand the relationship between lipoprotein metabolism and weight set-point.

DETAILED DESCRIPTION:
BACKGROUND:

The elevated high-density lipoprotein (HDL) cholesterol concentrations of long distance runners has been ascribed almost exclusively to increased muscle lipoprotein lipase. Based on data collected in cross-sectional and longitudinal studies, the investigators proposed an alternative theory: long-distance runners had the HDL-cholesterol metabolism of men who were below their sedentary weight rather than the HDL-cholesterol metabolism of lean sedentary men who were at their usual sedentary weight. In other analyses, they found that the most significant determinant of male runners' plasma HDL-cholesterol concentrations was the difference between the runners' greatest weight and their current weight. HDL- cholesterol levels were highest in runners who had lost the most weight, i.e., highest in those who were presumed to be the furthest below their weight set-point

The study was a result of a Program Announcement (PA) released in October, 1994 on Physical Activity and Cardiopulmonary Health. The PA was jointly sponsored by the NHLBI, the National Institute of Diabetes and Digestive and Kidney Diseases, and the National Institute of Nursing Research.

DESIGN NARRATIVE:

In this cross-sectional study, runners and sedentary men and women were measured for lipoprotein cholesterol, triglycerides, polyacrylamide gel electrophoresis of HDL and low-density lipoprotein subclasses, apolipoproteins A-I and B, intravenous fat clearance rate, post-heparin lipoprotein lipase and hepatic lipase, adipose tissue lipoprotein lipase, cholesteryl ester transfer activity, diet, percent body fat, and regional adiposity. It was hoped that the survey would confirm or reject the weight set-point hypothesis, provide a possible explanation of the lipoprotein differences between male and female runners, and elucidate the mechanism for the lipoprotein changes that occur during exercise-induced weight loss.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-05; Study Completion 1997-04 (Actual)

REFERENCES:
- [Background] Williams PT, Krauss RM. Associations of age, adiposity, menopause, and alcohol intake with low-density lipoprotein subclasses. Arterioscler Thromb Vasc Biol. 1997 Jun;17(6):1082-90. doi: 10.1161/01.atv.17.6.1082. PMID 9194758
- [Background] Williams PT. Deviations from maximum weight predict high-density lipoprotein cholesterol levels in runners: the National Runners' Health Study. Int J Obes Relat Metab Disord. 1997 Jan;21(1):6-13. doi: 10.1038/sj.ijo.0800352. PMID 9023594
- [Background] Williams PT. Evidence for the incompatibility of age-neutral overweight and age-neutral physical activity standards from runners. Am J Clin Nutr. 1997 May;65(5):1391-6. doi: 10.1093/ajcn/65.5.1391. PMID 9129467
- [Background] Williams PT, Dreon DM, Blanche PJ, Krauss RM. Variability of plasma HDL subclass concentrations in men and women over time. Arterioscler Thromb Vasc Biol. 1997 Apr;17(4):702-6. doi: 10.1161/01.atv.17.4.702. PMID 9108783
- [Background] Williams PT. Relationship of distance run per week to coronary heart disease risk factors in 8283 male runners. The National Runners' Health Study. Arch Intern Med. 1997 Jan 27;157(2):191-8. PMID 9009976
- [Background] Williams PT. High-density lipoprotein cholesterol and other risk factors for coronary heart disease in female runners. N Engl J Med. 1996 May 16;334(20):1298-303. doi: 10.1056/NEJM199605163342004. PMID 8609947